CLINICAL TRIAL: NCT04935281
Title: Percutaneous Repair of Acute Achilles Tendon Rupture With Assistance of Intraoperative Ultrasound: Does it Improves the Results of Repair?
Brief Title: Percutaneous Repair of Acute Achilles Tendon Rupture With Assistance of Intraoperative Ultrasound
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, ahmed m. samy, assisstant professor, Tanta University
Other Study IDs: Tanta H
Record Dates: First submitted 2021-05-27; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Acute Rupture of Achilles Tendon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- percutaneous repair with an intraoperative assissted ultrasound: a radiologist did an intraoperative ultrasound before the repair for identification the course of sural nerve and outline the medial and lateral edges of torn tendon.
  Interventions: Other: percutaneous repair with an intraoperative assisted ultrasound
- percutaneous repair without an intraoperative assissted ultrasound: the course of the sural nerve was determined according to the technique described by Blackmon et al .This technique depends on the leg length for location the point where the nerve crosses the lateral edge of the tendon
  Interventions: Other: percutaneous repair without an intraoperative assisted ultrasound

INTERVENTIONS:
Other: percutaneous repair with an intraoperative assisted ultrasound — Under general or regional anesthesia, the patient laid in prone position In group A, an intraoperative ultrasound was done by a radiologist before the repair .
  Groups: percutaneous repair with an intraoperative assissted ultrasound
Other: percutaneous repair without an intraoperative assisted ultrasound — For patients in group B, the course of the sural nerve was determined according to the technique described by Blackmon et al.The medial and lateral borders of both stumps were outlined by palpation with identification of the gap in-between. We used the technique described byMaffulli et al with six stab incisions, one cm each. Four incisions were on medial and lateral edge of the proximal stump and the other two were around distal stump.
  Groups: percutaneous repair without an intraoperative assissted ultrasound

SUMMARY:
This is a prospective randomized controlled study carried out between May 2016 and December 2020. It included 98 patients presented with acute rupture of Achilles tendon The patients were randomly distributed by closed envelop technique (49 in each group). Group A included those managed with the assistant of an intra-operative ultrasound. Group B included those done without ultrasound assistant

DETAILED DESCRIPTION:
A preoperative prophylactic dose of antibiotic was given intravenously in the form of 2gm of cephalosporin one hour before operation. Under general or regional anesthesia, the patient laid in prone position without a tourniquet and both feet out of the table for easily mobilization of the ankle joint. In group A, an intraoperative ultrasound was done by a radiologist before the repair for identification the course of sural nerve and outline the medial and lateral edges of torn tendon. Then ultrasound was repeated after repair for confirmation of adequate contact of both stumps and satisfactory strength of the repair by visualization of the tendon with passive motion of the ankle. For patients in group B, the course of the sural nerve was determined according to the technique described by Blackmon et al. This technique depends on the leg length for location the point where the nerve crosses the lateral edge of the tendon. The medial and lateral borders of both stumps were outlined by palpation with identification of the gap in-between. The technique of repair was standardized for all patients in both groups. We used the technique described by Maffulli et al

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50 years
* acute ( not more than two weeks) closed complete injury
* injury of Achilles tendon in zone 2 (the area between 3 and 6 cm from the insertion) according to Langergran and Lindholm

Exclusion Criteria:

* incomplete injury
* recurrent injury
* associated fracture ankle or foot
* previous history of local corticosteroids injection
* patients with neurovascular problem (e.g. diabetic, autoimmune …etc), smoking, and alcoholics

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: a prospective randomized control study
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
American Orthopedic Foot and An¬kle Society score | 4 years
  score from 0 to 100 with highest score is better
single leg rising | 3 years
  ability to stand on one leg
magnetic resonance image | one year
  assessment of healing of torn tendon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samy AM. Intra-operative ultrasound: does it improve the results of percutaneous repair of acute Achilles tendon rupture? Eur J Trauma Emerg Surg. 2022 Oct;48(5):4061-4068. doi: 10.1007/s00068-022-01926-x. Epub 2022 Mar 11. PMID 35275242